CLINICAL TRIAL: NCT00749372
Title: T2* Cardiac MRI Screening of Highly Transfused Patients With Myelodysplastic Syndrome
Brief Title: MRI Screening for Patients With Myelodysplastic Syndrome (MDS), Who Have Received Multiple Red Blood Cell Transfusions
Acronym: T2*MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 0803009687; CICL670A US23T
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Myelodysplastic Syndrome (MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes

ARMS (1):
- 1 (Other): Patients who meet eligibility will be sent for radiographic imaging to include T2* cardiac and liver MRI to ascertain quantification of organ-specific iron concentrations as well as cardiac left ventricular ejection fraction.
  Interventions: Other: T2* Cardiac and Liver MRI

INTERVENTIONS:
Other: T2* Cardiac and Liver MRI — Patients will undergo an MRI of the heart and liver.

SUMMARY:
A known risk of red blood cell transfusions is that it puts excess iron into the patient's body. Researchers are continually seeking the most effective method of measuring iron concentration. The purpose of this study is to determine how much iron has been deposited in a patient's heart and liver as a result of having received red blood cell transfusions using magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Male or Female patients will need documentation of diagnosis of Myelodysplastic Syndrome by previous bone marrow exam
* Male or female patients with MDS who have received at least 50 units of Red Blood Cell Transfusions.
* Serum ferritin > 1,000
* Written informed consent by the patient.

Exclusion Criteria:

* Contraindication to MRI, including cardiac pacemaker, brain aneurysm clip, implanted neurostimulator, insulin pump, cochlear implant, metal slivers in the eyes, intrauterine device or any other MRI incompatible metal implants or intractable claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-07-31 (Actual); Primary Completion 2013-03-29 (Actual); Study Completion 2013-03-29 (Actual)

PRIMARY OUTCOMES:
To evaluate the incidence of clinically significant cardiac iron overload in heavily transfused MDS patients using T2* MRI. | A single T2* MRI will be performed on eligible patients.

SECONDARY OUTCOMES:
Evaluate left ventricular ejection fraction as assessed by T2* MRI. | A single T2* MRI will be performed on eligible patients.
Evaluate liver iron concentration as assessed by R2* MRI | A single T2* MRI will be performed on eligible patients.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Feldman, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States